CLINICAL TRIAL: NCT04349644
Title: Enhancing Social Competence in Adults With Autism Spectrum Disorder: A Pilot RCT
Brief Title: Enhancing Social Competence in Adults With Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Blythe Corbett, Professor of Psychiatry and Behavioral Sciences, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 192271; 1R33MH120149-01A1 (NIH)
Record Dates: First submitted 2020-04-14; First posted 2020-04-16 (Actual); Results first posted 2025-03-07 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Autism Spectrum Disorder
Keywords: autism; social competence; theatre
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Social Skills

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SENSE Theatre (Experimental): A peer-mediated, theatre-based intervention designed to improve social cognition and behavior.
  Interventions: Behavioral: SENSE Theatre
- Waitlist Control Group (No Intervention): This group will not receive the intervention during the testing phase of the intervention but will eventually receive the theatre intervention.

INTERVENTIONS:
Behavioral: SENSE Theatre — A peer-mediated, theatre-based intervention that involves 10 sessions of approximately 3 hours each that culminates in a public performance.
  Arms: SENSE Theatre

SUMMARY:
SENSE Theatre®, combines several well-documented, effective behavioral strategies, such as the inclusion of trained peer models, theatre play techniques involving predictable (i.e., scripted) and flexible (improvised) role-play, and repeated performance of newly learned skills resulting in greater automaticity of behavior. The intervention has the potential to enhance social cognition and behavior in adults with autism spectrum disorder.

DETAILED DESCRIPTION:
Autism spectrum disorder (ASD) is characterized by primary impairment in social competence. Effects of current psychosocial interventions often fail to maintain or generalize and few employ rigorous experimental methods. Our treatment, SENSE Theatre®, combines several well-documented, effective behavioral strategies, such as the inclusion of trained peer models, theatre play techniques involving predictable (i.e., scripted) and flexible (improvised) role-play, and repeated performance of newly learned skills resulting in greater automaticity of behavior. Recent findings from a randomized control trial (RCT) show immediate between-group effects and evidence of target engagement on the hypothesized mechanism of action, memory for faces, which was evaluated by neuropsychological and event-related potential (ERP) measures. Moreover, the RCT demonstrated treatment effects on social communication skills that generalized to home and community settings. Finally, maintained treatment effects were observed on communication symptoms. The proposed project will extend these findings and provide a stronger test of efficacy using an RCT of SENSE Theatre with a sample of approximately 40 adult participants with ASD (18 to 35 years) randomized to experimental (EXP; N = 20) and a wait list control group (WLC; N = 20) in two separate cohorts. The RCT will assess target engagement of memory for faces and functional change in social interaction with peers using examiners blind to study treatment group assignment. The significance and size of treatment effects on these cognitive and behavioral outcomes will be measured using ANOVA and linear mixed models. Thus, the overarching aim of the study is to determine whether detected changes in face memory and social interaction are due to the SENSE Theatre® treatment and the extent to which these changes generalize and maintain. If predicted results occur, it will provide strong empirical support for a community-based treatment that has generalized effects on a set of core deficits that otherwise have life-long consequences for adults with ASD.

ELIGIBILITY:
ASD Inclusion Criteria:

* diagnosed with ASD based on DSM-V criteria (APA, 2013), by a psychologist, pediatrician or psychiatrist with expertise in ASD will be enrolled. ASD diagnosis will be corroborated by the Autism Diagnostic Observation Schedule (ADOS-2) (Lord, 2012).
* Only adults not currently supported by educational opportunities will be enrolled.
* Participants must have a full-scale IQ > or = 70 (WASI; (Wechsler, 2011))

ASD Exclusion Criteria:

* Adults with intellectual impairment (WASI; (Wechsler, 2011) score < 70.
* Participants with current, frequent and uncontrolled aggression toward other persons or property in the past 6 months will be excluded based on phone screening and questions from the Adult Behavior Checklist (Achenbach, 2001) (e.g., "Physically attacks people").
* Participants with evidence of suicidality based on care-provider report, self-report, or clinical interview (i.e., endorsement of suicidal ideation in the past month and/or suicidal behavior in the past three months on the Columbia Suicide Severity Rating Scale (Posner, 2011),
* Previous SENSE Theatre® participants will be excluded.

Care-giver Inclusion Criteria:

* must be at least 18 years of age
* must be a parent, close relative, or spouse of the adult participant with ASD.
* must be able to provide current and historical observations of the functioning of the participant with ASD.
* must live in close proximity to and have frequent contact with the participant with ASD.

Care-giver Exclusion Criteria:

- Anyone not meeting inclusion criteria.

Confederates Inclusion Criteria:

* must be at least 18 years of age
* typically developing individual with no neurodevelopmental disorder.
* must successfully complete training and demonstrate consistent administration of research protocols.

Confederate Exclusion Criteria:

- Anyone not meeting inclusion criteria.

Peers Inclusion Criteria:

* must be at least 18 years of age
* typically developing individual with no neurodevelopmental disorder.
* must have an expressed interest in supporting young adults and adults with developmental disabilities or ASD
* must successfully complete SENSE Theatre® training.

Peers Exclusion Criteria:

- Anyone not meeting inclusion criteria.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2025-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Blythe A Corbett, Ph.D., Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Corbett BA, Key AP, Klemencic ME, Muscatello RA, Jones D, Pilkington J, Burroughs C, Vandekar S. Investigating Social Competence in a Pilot Randomized Clinical Trial of a Theatre-Based Intervention Enhanced for Adults with Autism Spectrum Disorder. J Autism Dev Disord. 2025 Jan;55(1):130-146. doi: 10.1007/s10803-023-06214-0. Epub 2023 Dec 18. PMID 38109034

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Excluded (N=8). Not meeting inclusion criteria (N=5), Transportation issues (N=1), and unknown/reason not provided (N=2).
Period: Allocation/Pretest
Arm/Group | SENSE Theatre | Waitlist Control Group
Started | 29 | 35
Completed | 29 | 32
Not Completed | 0 | 3
Not completed — Lost to pretest | 0 | 3
Period: Posttest
Arm/Group | SENSE Theatre | Waitlist Control Group
Started | 29 | 32
Completed | 23 | 24
Not Completed | 6 | 8
Not completed — Lost to posttest | 0 | 8
Not completed — Discontinued intervention | 6 | 0
Period: Follow-up
Arm/Group | SENSE Theatre | Waitlist Control Group
Started | 23 | 24
Completed | 23 | 22
Not Completed | 0 | 2
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SENSE Theatre | Waitlist Control Group | Total
Number analyzed (Participants) | 29 | 35 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.48 (4.92) | 24.30 (5.97) | 24.38 (5.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 17 | 31
  Male | 15 | 18 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 27 | 34 | 61
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 22 | 26 | 48
  More than one race | 4 | 4 | 8
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 29 | 35 | 64
Autism Diagnostic Observation Schedule, 2nd Edition, Module 4 [Mean (Standard Deviation); unit: units on a scale] — The ADOS-2 is a semi-structured interview and series of activities to assess behaviors characteristic of autism spectrum disorder. The study focused on adults; therefore, we used Module 4. The scores are based on a diagnostic algorithm with scores ranging from 0 to 29. Higher scores indicate higher symptom severity.
  units on a scale | 7.34 (1.86) | 7.51 (1.62) | 7.43 (1.73)
Wechsler Abbreviated Scale of Intelligence, 2nd Edition [Mean (Standard Deviation); unit: units on a scale] — The WASI-2 is composed of four subtests: Block Design, Vocabulary, Matrix Reasoning and Similarities. The Full Scale IQ is derived from a summation of the subtests. The IQ Standard Score range is 40-160. Higher scores mean better outcomes.
  units on a scale | 102.45 (17.21) | 103.06 (22.86) | 102.78 (20.31)

OUTCOME MEASURES:

1. Primary Outcome: Change in Incidental Face Memory
Description: An event-related Potential Task that presents 51 novel faces and 51 novel houses one of each is randomly selected and presented 50 times (repeated). We are examining an increase in amplitude of 250-500 ms time window between the repeated and single face presentation. Positive values indicate better face memory.
Time Frame: Change from baseline to end of treatment (Week 11) and at Follow-up (Week 21)
Population: Number of participants analyzed at posttest. Two participants in SENSE Theatre and four in Waitlist Control had missing data. For follow-up the number of participants was SENSE Theatre N = 21 and Waitlist Control N = 20. Two participants in SENSE Theatre and two participants in Waitlist Control had missing data.
Measure: Mean (Standard Deviation); unit: microvolts
Arm/Group | SENSE Theatre | Waitlist Control Group
Number analyzed (Participants) | 21 | 20
microvolts
  Posttest (Week 11) | 0.6588 (0.9006) | -0.1604 (1.1751)
  Follow-up (Week 21) | 0.469 (1.279) | -0.77 (1.869)
Statistical Analysis 1: Comparison: SENSE Theatre vs Waitlist Control Group; Test type: Other — A series of Analysis of Covariance (ANCOVA) models were used to test the between-group differences on each dependent variable at the immediate posttest and at the follow-up periods separately using the pretest values as a covariate. Independent samples t-tests were used to identify statistically significant differences on all pretest dependent vari- ables; p = 0.016, ANCOVA; Posttest ANCOVA controlling for pretest values
Statistical Analysis 2: Comparison: SENSE Theatre vs Waitlist Control Group; Test type: Other — A series of Analysis of Covariance (ANCOVA) models were used to test the between-group differences on each depen- dent variable at the immediate posttest and at the follow-up periods separately using the pretest values as a covariate. Independent samples t-tests were used to identify statistically significant differences on all pretest dependent variables; p = 0.288, ANCOVA; Follow-up ANCOVA while controlling Pretest

2. Primary Outcome: Change in Contextual Assessment of Social Skills
Description: An observational assessment measure of social cognition and communication which includes two 3-minutes conversations with typically developing peers showing interested or bored demeanor. The behaviors are rated based on raw scores on a likert scale from 1 to 7 with 7 reflecting better ability. Only the Interested Condiiton was analyzed.
Time Frame: Change from baseline to end of treatment (Week 11) and at Follow-up (Week 21)
Population: Number of participants analyzed at posttest. One participant in Waitlist Control had missing data. For follow-up the number of participants was SENSE Theatre N = 23 and Waitlist Control N = 20. Two participants in Waitlist Control had missing data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SENSE Theatre | Waitlist Control Group
Number analyzed (Participants) | 23 | 23
units on a scale
  Vocal Expressiveness Posttest (Week 11) | 4.82 (1.708) | 4.52 (1.648)
  Quality of Rappport Posttest (Week 11) | 5.43 (1.409) | 5.13 (1.262)
  Vocal Expressiveness Follow-up (Week 21): number analyzed (Participants) | 23 | 20
  Vocal Expressiveness Follow-up (Week 21) | 4.30 (1.917) | 4.26 (1.485)
  Quality of Rapport Follow-up (Week 21): number analyzed (Participants) | 23 | 20
  Quality of Rapport Follow-up (Week 21) | 5.00 (1.168) | 4.85 (1.226)
Statistical Analysis 1: Comparison: SENSE Theatre vs Waitlist Control Group; Test type: Other — A series of Analysis of Covariance (ANCOVA) models were used to test the between-group differences on each dependent variable at the immediate posttest and at the follow-up periods separately using the pretest values as a covariate. Independent samples t-tests were used to identify statistically significant differences on all pretest dependent variables; p = 0.932, ANCOVA; Posttest ANCOVA controlling pretest value for CASS Vocal Expressiveness
Statistical Analysis 2: Comparison: SENSE Theatre vs Waitlist Control Group; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.221, ANCOVA; Posttest ANCOVA controlling for pretest for CASS Quality of Rapport
Statistical Analysis 3: Comparison: SENSE Theatre vs Waitlist Control Group; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.873, ANCOVA; Follow-up ANCOVA controlling for pretest Vocal Expressiveness
Statistical Analysis 4: Comparison: SENSE Theatre vs Waitlist Control Group; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.512, ANCOVA; Follow-up ANCOVA controlling for pretest Quality of Rapport

3. Primary Outcome: Change in Social Responsiveness Scale - Self (SRS)
Description: The SRS is a standardized measure of social competence self-administered by participants pertaining to behaviors characteristic of adults with ASD. T-scores range from scores of 38 to 90 with a mean of 50 and a standard deviation of 10. Higher scores reflect greater impairment. T-scores were used in the analyses. A decrease in scores from pretest to posttest or follow-up suggests a better outcome.
Time Frame: Change from baseline to end of treatment (Week 11) and at Follow-up (Week 21)
Population: Number of participants analyzed at posttest. One participant in SENSE Theatre had missing data. For follow-up the number of participants was SENSE Theatre N = 21 and Waitlist Control N = 22. Two participants in SENSE Theatre had missing data.
Measure: Mean (Standard Deviation); unit: T Scores
Arm/Group | SENSE Theatre | Waitlist Control Group
Number analyzed (Participants) | 22 | 24
T Scores
  Posttest (Week 11) | 63.23 (9.107) | 67.50 (10.338)
  Follow-up (Week 21): number analyzed (Participants) | 21 | 22
  Follow-up (Week 21) | 62.76 (10.183) | 65.77 (8.815)
Statistical Analysis 1: Comparison: SENSE Theatre vs Waitlist Control Group; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.05, ANCOVA; Posttest ANCOVA controlling for Pretest
Statistical Analysis 2: Comparison: SENSE Theatre vs Waitlist Control Group; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.393, ANCOVA; Follow-up ANCOVA controlling for Pretest

4. Primary Outcome: Change in Social Responsiveness Scale - Other (SRS)
Description: The SRS is a standardized measure of social competence administered by care-givers pertaining to behaviors characteristic of adults with ASD. T-scores range from scores of 38 to 90 with a mean of 50 and standard deviation of 10. Higher scores reflect greater impairment. T-scores were used in analyses. Decrease in scores from Pretest to Posttest or follow-up suggest better outcome.
Time Frame: Change from baseline to end of treatment (Week 11) and at Follow-up (Week 21)
Population: Number of participants analyzed at posttest. Two participants in Waitlist Control had missing data. For follow-up the number of participants was SENSE Theatre N = 20 and Waitlist Control N = 21. Three participants in SENSE Theatre and one in Waitlist Control had missing data.
Measure: Mean (Standard Deviation); unit: T Scores
Arm/Group | SENSE Theatre | Waitlist Control Group
Number analyzed (Participants) | 23 | 22
T Scores
  Posttest (Week 11) | 65.52 (9.853) | 66.23 (7.211)
  Follow-up (Week 21): number analyzed (Participants) | 20 | 21
  Follow-up (Week 21) | 63.95 (9.242) | 64.90 (8.282)
Statistical Analysis 1: Comparison: SENSE Theatre vs Waitlist Control Group; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.917, ANCOVA; Posttest ANCOVA controlling for pretest values
Statistical Analysis 2: Comparison: SENSE Theatre vs Waitlist Control Group; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.963, ANCOVA; Follow-up ANCOVA while controlling for pretest

5. Secondary Outcome: Cambridge Face Memory Test
Description: A standardized measure of face memory with 72 items. Total raw score ranges from 0-72. Any increase in the raw score pertaining to the number of faces identified constitutes an increase in face memory.
Time Frame: Change from baseline to end of treatment (Week 11) and at Follow-up (Week 21)
Population: Number of participants analyzed at posttest. One participant in SENSE Theatre had missing data. For follow-up the number of participants was SENSE Theatre N = 22 and Waitlist Control N = 21. One participant in SENSE Theatre and one participant in Waitlist Control had missing data.
Measure: Mean (Standard Deviation); unit: Raw score
Arm/Group | SENSE Theatre | Waitlist Control Group
Number analyzed (Participants) | 22 | 24
Raw score
  Posttest (Week 11) | 47.5 (10.796) | 45.75 (8.936)
  Follow-up (Week 21): number analyzed (Participants) | 22 | 21
  Follow-up (Week 21) | 47.68 (13.375) | 49.24 (9.060)
Statistical Analysis 1: Comparison: SENSE Theatre vs Waitlist Control Group; Test type: Other — A series of Analysis of Covariance (ANCOVA) models were used to test the between-group differences on each dependent variable at the immediate posttest (Week 11) and at the follow-up (Week 21) periods separately using the pretest values as a covariate; p = 0.879, ANCOVA; Posttest ANCOVA controlling pretest
Statistical Analysis 2: Comparison: SENSE Theatre vs Waitlist Control Group; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.216, ANCOVA; Follow-up ANCOVA controlling for pretest

6. Secondary Outcome: Wechsler Memory Scale Face Memory Delay Test
Description: A standardized measure of face memory in which the participant is exposed to 24 faces in which they must remember amidst an array of 48 faces presented after a 30-minute delay. Raw scores range from 0-48 and are converted to age-adjusted scaled scores ranging from 1 to 19 (Mean of 10 and standard deviation of 3). Higher scaled scores reflect better delayed face memory. Scaled scores were used for analyses.
Time Frame: Change from baseline to end of treatment (Week 11) and at Follow-up (Week 21)
Population: Number of participants analyzed at posttest. For follow-up the number of participants was SENSE Theatre N = 23 and Waitlist Control N = 22.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SENSE Theatre | Waitlist Control Group
Number analyzed (Participants) | 23 | 24
units on a scale
  Posttest (Week 11) | 8.35 (3.242) | 7.88 (2.740)
  Follow-up (Week 21): number analyzed (Participants) | 23 | 22
  Follow-up (Week 21) | 8.35 (4.052) | 8.05 (3.184)
Statistical Analysis 1: Comparison: SENSE Theatre vs Waitlist Control Group; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.166, ANCOVA; Posttest ANCOVA controlling for pretest
Statistical Analysis 2: Comparison: SENSE Theatre vs Waitlist Control Group; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.331, ANCOVA; Follow-up ANCOVA controlling for pretest

7. Secondary Outcome: Wechsler Memory Scale Face Memory Test
Description: A standardized measure of face memory in which the participant is exposed to 24 faces in which they must remember amidst an array of 48 faces presented immediately. Raw scores range from 0-48 and are converted to age-adjusted scaled scores ranging from 1 to 19 (Mean of 10 and standard deviation of 3). Higher scaled scores reflect better face memory. Scaled scores were used for analyses.
Time Frame: Change from baseline to end of treatment (Week 11) and at Follow-up (Week 21)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SENSE Theatre | Waitlist Control Group
Number analyzed (Participants) | 23 | 24
units on a scale
  Posttest (Week 11) | 8.13 (3.507) | 7.67 (2.914)
  Follow-up (Week 21): number analyzed (Participants) | 23 | 22
  Follow-up (Week 21) | 8.17 (3.927) | 8.50 (2.972)
Statistical Analysis 1: Comparison: SENSE Theatre vs Waitlist Control Group; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.507, ANCOVA; Posttest controlling for pretest
Statistical Analysis 2: Comparison: SENSE Theatre vs Waitlist Control Group; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.064, ANCOVA; Follow-up controlling for pretest

8. Secondary Outcome: Adaptive Behavior Assessment System (ABAS) - Self-Report Global Adaptive Composite
Description: The ABAS measures adaptive living skills, completed via self-administration, using a Standardized Scale in which in which scores ranging from ~70 to ~120, with 85 to 115 reflecting the broad average range. Lower scores represent greater impairment.
Time Frame: Change from baseline to end of treatment (Week 11) and at Follow-up (Week 21)
Population: Number of participants analyzed at posttest. For follow-up the number of participants was SENSE Theatre N = 21 and Waitlist Control N = 21. Two participants in SENSE Theatre and one participant in Waitlist Control had missing data.
Measure: Mean (Standard Deviation); unit: Standard Score
Arm/Group | SENSE Theatre | Waitlist Control Group
Number analyzed (Participants) | 23 | 24
Standard Score
  Posttest (Week 11) | 89.04 (16.328) | 85.83 (19.175)
  Follow-up (Week 21): number analyzed (Participants) | 21 | 21
  Follow-up (Week 21) | 88.57 (12.651) | 87.14 (15.907)
Statistical Analysis 1: Comparison: SENSE Theatre vs Waitlist Control Group; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.706, ANCOVA; Posttest controlling for pretest
Statistical Analysis 2: Comparison: SENSE Theatre vs Waitlist Control Group; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.987, ANCOVA; Follow-up ANCOVA controlling for pretest

9. Secondary Outcome: Adaptive Behavior Assessment System (ABAS) - Other-Report Global Adaptive Composite
Description: The ABAS measures adaptive living skills, completed by a caregiver or partner, using a Standardized Scale in which scores ranging from ~70 to ~120, with 85 to 115 reflecting the broad average range. Lower scores represent greater impairment.
Time Frame: Change from baseline to end of treatment (Week 11) and at Follow-up (Week 21)
Population: Number of participants analyzed at posttest. Two participants in Waitlist Control had missing data. For follow-up the number of participants was SENSE Theatre N = 20 and Waitlist Control N = 21. Three participants in SENSE Theatre and one participant in Waitlist Control had missing data.
Measure: Mean (Standard Deviation); unit: Standard Score
Arm/Group | SENSE Theatre | Waitlist Control Group
Number analyzed (Participants) | 23 | 22
Standard Score
  Posttest (Week 11) | 76.61 (13.313) | 79.73 (15.761)
  Follow-up (Week 21): number analyzed (Participants) | 20 | 21
  Follow-up (Week 21) | 77.20 (11.372) | 78.90 (16.435)
Statistical Analysis 1: Comparison: SENSE Theatre vs Waitlist Control Group; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.475, ANCOVA; Posttest ANCOVA controlling for pretest
Statistical Analysis 2: Comparison: SENSE Theatre vs Waitlist Control Group; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.668, ANCOVA; Follow-up ANCOVA controlling for pretest

10. Secondary Outcome: State-Trait Anxiety Inventory (STAI) Scale
Description: The STAI is a measure of current (State) and enduring (Trait) anxiety that is completed by the participant. There are 20 items for each domain on a 4-point scale (1 = Almost Never, 4 = Almost Always). Scores range from 20 to 80, with higher scores reflecting greater anxiety.
Time Frame: Change from baseline to end of treatment (Week 11) and at Follow-up (Week 21)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Raw score
Arm/Group | SENSE Theatre | Waitlist Control Group
Number analyzed (Participants) | 23 | 24
Raw score
  State Posttest (Week 11) | 39.13 (8.498) | 42.42 (12.058)
  Trait Posttest (Week 11) | 42.43 (9.539) | 48.13 (4.266)
  State Follow-up (Week 21): number analyzed (Participants) | 23 | 22
  State Follow-up (Week 21) | 39.57 (10.854) | 41.00 (12.585)
  Trait Follow-up (Week 21): number analyzed (Participants) | 23 | 22
  Trait Follow-up (Week 21) | 42.83 (9.731) | 47.86 (13.892)
Statistical Analysis 1: Comparison: SENSE Theatre vs Waitlist Control Group; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.525, ANCOVA; Posttest ANCOVA controlling for pretest for STAI STATE
Statistical Analysis 2: Comparison: SENSE Theatre vs Waitlist Control Group; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.307, ANCOVA; Posttest ANCOVA controlling for pretest for STAI Trait
Statistical Analysis 3: Comparison: SENSE Theatre vs Waitlist Control Group; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.950, ANCOVA; Follow-up ANCOVA controlling for pretest for STAI State
Statistical Analysis 4: Comparison: SENSE Theatre vs Waitlist Control Group; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.459, ANCOVA; Follow-up ANCOVA controlling for pretest for STAI Trait

11. Secondary Outcome: The Adult Self Report (ASR)
Description: The ASR is a 126-item self-report questionnaire assessing aspects of emotional health. T scores range from 40 to 100 with a mean of 50 and a standard deviation of 10. The primary variables of interest were Depressive Problems and Anxiety Problems. Higher scores indicate more depressive or anxiety problems. A T score of 70 or higher is considered clinically significant.
Time Frame: Change from baseline to end of treatment (Week 11) and at Follow-up (Week 21)
Population: Number of participants analyzed at posttest. One participant in Waitlist Control had missing data. For follow-up the number of participants was SENSE Theatre N = 21 and Waitlist Control N = 22. Two participants in SENSE Theatre had missing data.
Measure: Mean (Standard Deviation); unit: T Scores
Arm/Group | SENSE Theatre | Waitlist Control Group
Number analyzed (Participants) | 23 | 23
T Scores
  Depression problems Posttest (Week 11) | 60.83 (10.347) | 63.39 (11.555)
  Anxiety Problems Posttest (Week 11) | 53.83 (6.485) | 59.00 (8.650)
  Depression problems Follow-up (Week 21): number analyzed (Participants) | 21 | 22
  Depression problems Follow-up (Week 21) | 59.86 (10.744) | 62.68 (10.191)
  Anxiety problems Follow-up (Week 21): number analyzed (Participants) | 21 | 22
  Anxiety problems Follow-up (Week 21) | 56.19 (8.744) | 60.27 (10.161)
Statistical Analysis 1: Comparison: SENSE Theatre vs Waitlist Control Group; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.215, ANCOVA; Posttest ANCOVA controlling for pretest for Depression problems
Statistical Analysis 2: Comparison: SENSE Theatre vs Waitlist Control Group; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.093, ANCOVA; Posttest ANCOVA controlling for pretest for Anxiety problems
Statistical Analysis 3: Comparison: SENSE Theatre vs Waitlist Control Group; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.223, ANCOVA; Follow-up ANCOVA controlling for pretest for Depression problems
Statistical Analysis 4: Comparison: SENSE Theatre vs Waitlist Control Group; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.838, ANCOVA; Follow-up ANCOVA controlling for pretest for Anxiety problems

12. Secondary Outcome: The Adult Behavior Checklist (ABCL)
Description: The ABCL is a 126-item caregiver-report questionnaire assessing aspects of emotional health. T scores range from 40 to 100 with a mean of 50 and a standard deviation of 10. The primary variables of interest were Depressive Problems and Anxiety Problems. Higher scores indicate more depressive or anxiety problems. A T score of 70 or higher is considered clinically significant.
Time Frame: Change from baseline to end of treatment (Week 11) and at Follow-up (Week 21)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: T Scores
Arm/Group | SENSE Theatre | Waitlist Control Group
Number analyzed (Participants) | 23 | 22
T Scores
  Depression problems posttest (week 11) | 61.26 (9.314) | 63.91 (10.099)
  Anxiety problems posttest (week 11) | 58.13 (9.411) | 60.36 (8.644)
  Depression problems follow-up (week 21): number analyzed (Participants) | 20 | 21
  Depression problems follow-up (week 21) | 60.25 (9.962) | 64.00 (9.327)
  Anxiety problems follow-up (week 21): number analyzed (Participants) | 20 | 21
  Anxiety problems follow-up (week 21) | 58.90 (9.978) | 61.43 (8.483)
Statistical Analysis 1: Comparison: SENSE Theatre vs Waitlist Control Group; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.716, ANCOVA; Posttest ANCOVA controlling for pretest Depressive problems
Statistical Analysis 2: Comparison: SENSE Theatre vs Waitlist Control Group; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.214, ANCOVA; Posttest ANCOVA controlling for pretest Anxiety problems
Statistical Analysis 3: Comparison: SENSE Theatre vs Waitlist Control Group; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.983, ANCOVA; Follow-up ANCOVA controlling for pretest Depressive problems
Statistical Analysis 4: Comparison: SENSE Theatre vs Waitlist Control Group; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 0.454, ANCOVA; Follow-up ANCOVA controlling for pretest for Anxiety problems

ADVERSE EVENTS:
Time Frame: Baseline through study completion (on average, approximately 18 weeks).
Arm/Group | SENSE Theatre | Waitlist Control Group
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/35
Other Adverse Events (participants affected / at risk) | 0/29 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-07-19): https://cdn.clinicaltrials.gov/large-docs/44/NCT04349644/Prot_001.pdf
  • Statistical Analysis Plan (2019-04-26): https://cdn.clinicaltrials.gov/large-docs/44/NCT04349644/SAP_002.pdf
  • Informed Consent Form (2020-01-16): https://cdn.clinicaltrials.gov/large-docs/44/NCT04349644/ICF_000.pdf